CLINICAL TRIAL: NCT03260634
Title: The Study of Voriconazole Trough Level in the First Two Weeks After Administration in King Chulalongkorn Memorial Hospital.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Other Study IDs: 496-59
Record Dates: First submitted 2017-08-08; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-01

CONDITIONS: Voriconazole; Fungal Infection
Keywords: voriconazole; therapeutic drug monitoring
MeSH Terms: conditions — Mycoses | interventions — Voriconazole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Voriconazole: Patient was received voriconazole according to individual indication. The starting dose is 6 mg/kg iv twice daily for two dosages, followed by 4 mg/kg iv twice daily in intravenous form or a loading dose of 400 mg twice daily for two doses is used (for individuals >40 kg), followed by 200 mg twice daily, and in individuals <40 kg the maintenance dose is 100 mg twice daily in oral form.
  The dosage was adjusted by drug level and toxicity. The duration of drug used was depended on indication of treatment.
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole

SUMMARY:
Invasive fungal infections are a significant cause of morbidity and mortality in immunocompromised host such as prolong neutropenic patients , post transplantation patients, malignancies or advanced AIDS . The majority of these infections were caused by Aspergillus species, which the first line of treatment is antifungal agent, Voriconazole , a triazole antifungal drug which was approved by the Food and Drug Administration in May 2002 for the treatment of invasive aspergillosis and refractory infections of Scedosporium apiospermum and Fusarium spp. There are two forms of Voriconazole , oral and intravenous form. The recommendation dose is 6 mg/kg twice daily for two dosages, followed by 4 mg/kg twice daily in intravenous form or a loading dose of 400 mg twice daily for two doses is used (for individuals >40 kg), followed by 200 mg twice daily, and in individuals <40 kg the maintenance dose is 100 mg twice daily in oral form.

Voriconazole has a narrow therapeutic window and nonlinear pharmacokinetic profile with wide inter-individual and intra-individual variability, such as age, race, genotypic variation, liver dysfunction, the presence of food and drug-drug interactions with CYP450 inhibitors. These large variations in pharmacokinetics may be associated with decreased efficacy or increased toxicity. Therefore , monitoring of serum trough concentrations is recommended in the following infections: invasive aspergillosis treatment , endophthalmitis; meningitis or osteoarticular infections due to Exserohilum rostratum.

In Thai population , there are different genetic polymorphism from Caucasian ,resulting in a different response to the initial dose and there is limited resources in Thailand , mostly patients are unaccessible for Voriconazole level. Especially,in the period of starting drug, which is the critical period for patients ,most of them are post chemotherapy which may have gastrointestinal problems, mucositis , vomiting or diarrhea ,as well as receiving multiple concurrent medications. All of these affect drug absorption,drug level and efficacy of treatment. Thus, this study was designed to evaluated Voriconazole level in Thai patients in the first two week after administration.

Primary question

* From the first collected of Voriconazole drug level , Are the invasive fungal infection patients in King Chulalongkorn Memorial Hospital achieved the drug level more than 60% ?

Secondary question

* Which factor affecting Voriconazole through level in the first two weeks after administration?

Research Design

* Observational Studies (Descriptive retrospective and prospective study)

Research Methodology

Target Population

* Patients received Voriconazole for treatment or prophylaxis invasive fungal infection

Study population

* Patients in King Chulalongkorn Memorial hospital received Voriconazole for treatment or prophylaxis invasive fungal infection

Sample size

n= ZZ/2P(1-P) /dd

* n = sample size
* P =Incident rate
* From the pilot study of 15 Invasive fungal infection patients in King Chulalongkorn memorial hospital from February to September 2015 , 60% ( 9 of 15 patients) of the first collected of Voriconazole trough level achieved the therapeutic level.

replaced P = 0.6

* Z = 95% confident interval = 1.96
* d = acceptable error = 0.10

n = (1.96) (1.96) (0.60)(1-0.60) / (0.10)(0.10)

n =92 , sample size = 92

Study processing and data collection

Data collection

* Collected data of patients received Voriconazole in first two weeks of treatment or prophylaxis invasive fungal infection in King Chulalongkorn Memorial hospital in 2015-2017 from outpatient records , inpatient records and computer database in King Chulalongkorn Memorial hospital. This data included
* Baseline characteristics : sex, age ,weight ,BMI ,co-morbid ,personal history of smoking or alcohol drinking
* Basic laboratory investigation : complete blood count , Creatinin , liver function test , albumin level
* Gastrointestinal problems
* Indication of Voriconazole treatment
* Data of invasive fungal infection :
* Data of Voriconazole usage : Loading dose, Maintenance dose, Trough level , Data of drug adjustment, Concurrent medication used, Side effect
* All data was summarized and recorded in case report forms.

Data Analysis and Statistics

The data was analysed by computer using SPSS17 program This study used descriptive statistics ,describing general information, age, results, laboratory results and side effects of the drug in mean ,percentage or standard deviation. And used the chi-square test for analysis of the proportion of patients with serum drug levels within the therapeutic range.

This study used a confidence level of 95%, p-value less than 0.05 was statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Thai patient in King Chulalongkorn Memorial Hospital , age between 18 and 80 years old
* Receiving Voriconazole for treatment or prophylaxis invasive fungal infection

Exclusion Criteria:

* Severe hepatic or renal dysfunction
* Pregnancy
* Presence of history of allergy to any Azole antifungal agents
* Death within 2 weeks after treatment of invasive fungal infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thai patient in King Chulalongkorn Memorial Hospital ,Bangkok , Thailand, age between 18 and 80 year olds ,receiving Voriconazole for treatment or prophylaxis invasive fungal infection , between 2015-2017.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-10-01 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieved therapeutic level of voriconazole in the first two weeks after administration | 2015-2017

SECONDARY OUTCOMES:
Factors have significant impact to voriconazole through level . | 2015-2017
  Factors that have significant impact to voriconazole through level will be assess in this study such as drug interaction , oral mucositis .

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn university, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamada Y, Tokimatsu I, Mikamo H, Kimura M, Seki M, Takakura S, Ohmagari N, Takahashi Y, Kasahara K, Matsumoto K, Okada K, Igarashi M, Kobayashi M, Mochizuki T, Nishi Y, Tanigawara Y, Kimura T, Takesue Y. Practice guidelines for therapeutic drug monitoring of voriconazole: a consensus review of the Japanese Society of Chemotherapy and the Japanese Society of Therapeutic Drug Monitoring. J Infect Chemother. 2013 Jun;19(3):381-92. doi: 10.1007/s10156-013-0607-8. Epub 2013 May 15. No abstract available. PMID 23673473
- [Background] Park WB, Kim NH, Kim KH, Lee SH, Nam WS, Yoon SH, Song KH, Choe PG, Kim NJ, Jang IJ, Oh MD, Yu KS. The effect of therapeutic drug monitoring on safety and efficacy of voriconazole in invasive fungal infections: a randomized controlled trial. Clin Infect Dis. 2012 Oct;55(8):1080-7. doi: 10.1093/cid/cis599. Epub 2012 Jul 3. PMID 22761409
- [Background] Pascual A, Calandra T, Bolay S, Buclin T, Bille J, Marchetti O. Voriconazole therapeutic drug monitoring in patients with invasive mycoses improves efficacy and safety outcomes. Clin Infect Dis. 2008 Jan 15;46(2):201-11. doi: 10.1086/524669. PMID 18171251
- [Background] Tan K, Brayshaw N, Tomaszewski K, Troke P, Wood N. Investigation of the potential relationships between plasma voriconazole concentrations and visual adverse events or liver function test abnormalities. J Clin Pharmacol. 2006 Feb;46(2):235-43. doi: 10.1177/0091270005283837. PMID 16432276
- [Background] Ueda K, Nannya Y, Kumano K, Hangaishi A, Takahashi T, Imai Y, Kurokawa M. Monitoring trough concentration of voriconazole is important to ensure successful antifungal therapy and to avoid hepatic damage in patients with hematological disorders. Int J Hematol. 2009 Jun;89(5):592-9. doi: 10.1007/s12185-009-0296-3. Epub 2009 Apr 2. PMID 19340528
- [Background] Patterson TF, Thompson GR 3rd, Denning DW, Fishman JA, Hadley S, Herbrecht R, Kontoyiannis DP, Marr KA, Morrison VA, Nguyen MH, Segal BH, Steinbach WJ, Stevens DA, Walsh TJ, Wingard JR, Young JA, Bennett JE. Practice Guidelines for the Diagnosis and Management of Aspergillosis: 2016 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2016 Aug 15;63(4):e1-e60. doi: 10.1093/cid/ciw326. Epub 2016 Jun 29. PMID 27365388